CLINICAL TRIAL: NCT02967588
Title: Development and Feasibility of a Brief Hospital-Based Intervention to Support Medication Adherence Following Acute Coronary Syndrome
Brief Title: An Intervention to Support Medication Adherence Following Acute Coronary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: v1 06-09-16
Record Dates: First submitted 2016-10-11; First posted 2016-11-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2016-09

CONDITIONS: Acute Coronary Syndrome
Keywords: Medication adherence; Behavioural intervention; Acute coronary syndrome; Medication beliefs; Implementation intentions
MeSH Terms: conditions — Acute Coronary Syndrome; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Behavioral: Intervention group

INTERVENTIONS:
Behavioral: Intervention group — All stages of the intervention will take place during hospitalization. Patients will complete a questionnaire about their personal beliefs about medicines. Patients responses to this questionnaire will form the basis of Session 1 where beliefs about medicines will be discussed. Any negative beliefs or concerns will be discussed and beliefs about drug necessity will be encouraged.
  Session 2 will focus on developing specific action plans for taking medication at home. Patients will be asked to formulate an if-then plan ('If it is time X in place Y and I am doing Z, then I will take my pill dose').
  Prior to discharge, patients will complete the beliefs questionnaire again to see if there has been any shift in their beliefs about medications. Patients will also be asked to provide detailed feedback about the study. The investigators want to know whether the intervention setting, timing, content and delivery method seem to be acceptable to patients.

SUMMARY:
Background Medication adherence following acute coronary syndrome (ACS) is often sub-optimal and is associated with poor clinical outcomes. Non-adherence can be considered intentional or unintentional. Findings ways to improve adherence is an important area of research with widespread clinical implications, however, previous interventions have generally been ineffective. The investigators propose an intervention that challenges both intentional and unintentional non-adherence in patients hospitalised following ACS.

Objectives The objective of this study is to determine the feasibility of a hospital-based intervention aimed at supporting medication adherence in patients following an ACS.

Methods Patients admitted to hospital with an ACS will be recruited for this study. The study will target both intentional and unintentional non-adherence over two sessions through challenging treatment beliefs and formulating specific action plans to encourage habit formation. Patients will be asked to provide in-depth feedback around the acceptability of the intervention. As this is a feasibility study, outcomes (i.e. medication adherence) will not be collected.

Dissemination If this study seems to be practical to deliver and acceptable to patients then it will inform the design of a future randomized-controlled pilot study to test the effectiveness of the intervention delivered by hospital pharmacists on a study outcome (i.e. medication adherence).

DETAILED DESCRIPTION:
Intervention details

* All stages of the intervention will take place during hospitalization.
* Firstly, patients will complete a questionnaire based on the Beliefs about Medication Questionnaire-Specific (BMQ-S) (Horne & Weinmen, 1999).
* Patients responses to this questionnaire will form the basis of Session 1 where beliefs about medicines will be discussed. The aim is to identify any negative or erroneous beliefs patients have that may prevent them from taking their medicines after they leave the hospital.
* Session 2 will focus on developing specific action plans for taking medication at home. Patients will be asked to formulate an if-then plan ('If it is time X in place Y and I am doing Z, then I will take my pill dose'. The aim is to make taking their medicines as much a part of their daily routine as possible.
* Prior to discharge, patients will complete the beliefs questionnaire again to see if there has been any shift in their beliefs about medications.
* Patients will also be asked to provide detailed feedback about the study. The investigators want to know whether the intervention setting (i.e. hospital-based), timing (i.e. straight after an ACS), content (i.e. targeting both intentional and unintentional non-adherence) and interventionist (i.e. PhD candidate) seem to be acceptable to patients.
* Feedback will be gathered after completion of the intervention and also during a follow up phone call 2-3 weeks after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ACS
* ACS primary reason for hospitalization
* Patients to be prescribed medications for secondary prevention (i.e. antiplatelet drugs, statins, ACEi, ARBs, β-blockers)
* Sufficient spoken English to participate in the study

Exclusion Criteria:

* Developed ACS as a secondary condition (i.e. perioperative MI)
* Not prescribed medications for secondary prevention (i.e. antiplatelet drugs, statins, ACEi, ARBs, β-blockers)
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Treatment beliefs | During index hospitalisation, within two days of admission.
  Beliefs about medications will be compared pre-post intervention using responses from the BMQ-S, Separate necessity and concerns scores will be calculated (5-items each, total scores ranging 5-25) along with the BMQ differential (necessity score - concerns score) (Gujral et al., 2014).

SECONDARY OUTCOMES:
Initial patient study feedback | During index hospitalisation, within two days of admission.
  Patients will complete a study feedback questionnaire which will determine its acceptability to patients (setting, timing, content, delivery method).
Detailed patient study feedback | Within three weeks post-discharge
  Detailed patient feedback will be gathered 2-3 weeks after discharge via a phone call. A brief semi-structured interview will be undertaken and study acceptability will be assessed (setting, timing, content, delivery method). The follow up call will be audio recorded, transcribed and used to evaluate the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No